CLINICAL TRIAL: NCT05953064
Title: Effects of DHA-NAT on Postprandial Lipidaemia in Healthy Male Subjects (FEAST): a Randomised, Double-blind, Placebocontrolled, Crossover Study
Brief Title: Effects of DHA-NAT on Postprandial Lipidaemia in Healthy Male Subjects
Acronym: FEAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Principal Investigator, Clinical Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FEAST
Record Dates: First submitted 2023-06-20; First posted 2023-07-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-11

CONDITIONS: Hypertriglyceridemia
Keywords: N-acyl taurine
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DHA-NAT (Experimental): Oral administration with a test meal of 55 kJ/kg bodyweight, with 60% of calories from fat.
  Interventions: Other: DHA-NAT
- Placebo (Placebo Comparator): Oral administration with a test meal of 55 kJ/kg bodyweight, with 60% of calories from fat.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: DHA-NAT — Endogenous metabolite of omega-3 fatty acid docosahexaenoic acid
  Other Names: C22:6 N-acyl taurine
  Arms: DHA-NAT
Other: Placebo — Vehicle control (H2O) for the intervention used in the experimental arm (DHA-NAT).
  Arms: Placebo

SUMMARY:
This study is an investigator-initiated, randomised, double-blind, placebo-controlled, cross-over human trial investigating the effect of DHA-NAT (C22:6 N-acyl taurine, an endogenous metabolite derived from the omega-3 fatty acid, docosahexaenoic acid) on postprandial plasma triglyceride levels following a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Age between 18 and 30 years
* Body mass index between 18.5-25 kg/m2
* Informed consent
* Moderate level of physical activity assessed with IPAQ (short version)

Exclusion Criteria:

* Use of fish-oil/omega-3 FA supplements within the last 3 months
* Regular tobacco smoking or use of other nicotine-containing products
* Allergy or intolerance to ingredients included in the standardised meals
* Weekly intake of fish >350 g (23)
* First-degree relatives with diabetes and/or glycated haemoglobin (HbA1c) >48 mmol/mol, familial hypercholesterolemia/hyperlipidemia
* Anaemia (haemoglobin below 8.3 mmol/L)
* Alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) >2 times upper normal values (Normal values: ALAT < 70 U/L, ASAT <45 U/L)
* Nephropathy (serum creatinine >105 μmol/L) and/or albuminuria (>30 mg/g albumin in urine))
* History of hepatobiliary or gastrointestinal disorder(s)
* Any physical or psychological condition, or ongoing medication, that the investigator evaluates would interfere with trial participation, including any acute or chronic illnesses

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Plasma triglyceride | 0-240 minutes
  Change in incremental area-under-curve plasma triglyceride

SECONDARY OUTCOMES:
Plasma GLP-1 | 0-240 minutes
  Plasma GLP-1 profile
Plasma N-acyl taurine species | 0-240 minutes
  Profile of plasma n-acyl taurine species
Plasma ApoB48 | 0-240 minutes
  Plasma ApoB48 profile
Satiety, hunger and appetite | 0-240 minutes
  Development during study day recorded by visual analogue scale (VAS), 0-10 cm where 0 = not in agreement with statement and 10 = in agreement with statement.
Food intake (g) | t=240 minutes
  Grams consumed of a standard ad libitum meal
Food intake (kcal) | t=240 minutes
  kcal consumed of a standard ad libitum meal
Plasma triglyceride (TG) distribution | 0-240 minutes
  total TG, and TG in HDL, LDL and VLDL cholesterol, remnant TG
Plasma free fatty acid species | 0-240 minutes
  Total fatty acids profile
Plasma cholesterol | 0-240 minutes
  Total cholesterol, HDL, LDL, VLDL, remnant cholesterol
Plasma level of glucose regulating hormones | 0-240 minutes
  Insulin, glucagon and gastric inhibitory polypeptide
Plasma amino acids | 0-240 minutes
  Total amino acids profile
Plasma glucose | 0-240 minutes
  Plasma glucose profile
Plasma bile acid species | 0-240 minutes
  Plasma bile acid profile
Gall bladder emptying: Cholecystokinin | 0-240 minutes
  Cholecystokinin profile
Gall bladder emptying: Ultrasonography | 0-240 minutes
  Difference in volume from most to least full
Gastric emptying: Paracetamol | 0-240 minutes
  Plasma acetaminphen profile
Stool quality | Up to 24 hours from ingestion of test meal or until first bowel movement if later than 24 hours.
  Self-assessment of stool quality by the Bristol Stool Scale (1-7, where 1 = most solid and 7 = least solid)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Herlev-Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No